CLINICAL TRIAL: NCT03633565
Title: A Comparative Study of Strategies for Management of Duchenne Myopathy in Assiut University Children Hospital
Brief Title: Comparative Study of Strategies for Management of Duchenne Myopathy (DM)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Nancy Alaa, principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: smdmauch
Record Dates: First submitted 2018-08-12; First posted 2018-08-16 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Myopathy
MeSH Terms: conditions — Muscular Diseases | interventions — Sildenafil Citrate; Phosphodiesterase Inhibitors; Prednisolone; Steroids; Mesenchymal Stem Cell Transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Steroid (Active Comparator): prednisolone 20 mg tablet by mouth taken once daily for 10 days each month for 2 years
  Interventions: Drug: Prednisolone (Steroids)
- Phosphodiestrase inhibitors (Active Comparator): sildenafil 25 mg tablet by mouth once daily for 2 years
  Interventions: Drug: Sildenafil (Phosphodiesterase inhibitors)
- Mesenchymal stem cell transplantation (Experimental): The cells can be injected intramuscular in several points in the muscle alternatively they can be injected in the motor point of the muscle. A motor point is the point at which the motor branch of the innervating nerve enters the muscle). This injection is repeated every 6 month up to 2 years.
  Interventions: Procedure: Mesenchymal stem cell transplantation

INTERVENTIONS:
Drug: Sildenafil (Phosphodiesterase inhibitors) — tablet 25mg
  Other Names: sildenafil; viagra
  Arms: Phosphodiestrase inhibitors
Drug: Prednisolone (Steroids) — tablet 20 mg
  Other Names: Prednisolone 20 mg
  Arms: Steroid
Procedure: Mesenchymal stem cell transplantation — stem cell transplantation intramuscular
  Arms: Mesenchymal stem cell transplantation

SUMMARY:
1. Comparing different lines of treatment of Duchenne Myopathy (DM) and assessment of new lines of treatment (mesenchymal stem cell, phosphodiesterase inhibitors) in reducing the impact of disability in the patients with Duchenne Myopathy and slowing the progression of cardiomyopathy
2. Upsetting and implementation of the best treatment plan for those children with Duchenne myopathy which is suitable for the available resources in Assiut University Children Hospital

DETAILED DESCRIPTION:
Duchenne muscular dystrophy(DMD) is the most commonly inherited pediatric muscular disorder. It is an X-linked genetic progressive and degenerative myopathy characterized by progressive weakness, which can lead to loss of motor functions in puberty as well as cardiac,respiratory involvement and premature death. The disease is one of a group of myopathies that differ depending on the degree of severity and the affected muscle types. It occurs at a rate of approximately 1:3500 male births and arises due to spontaneous mutations in the Dystrophin gene (locus Xp21.2); 65% of causative mutations are intragenic deletions, 6-10% are intragenic duplications and 30-35% are point mutations (along with other sequence variations). The disease is caused by a deficiency of Dystrophin or the synthesis of functionally impotent Dystrophin, a critical protein component of the Dystrophin glycoprotein complex acting as a link between the cytoskeleton and the extracellular matrix in skeletal and cardiac muscles. A consequence of Dystrophin glycoprotein complex inefficiency is muscle fragility, contraction-induced damage, necrosis and inflammation.

Glucocorticoid can prolong ambulation by 2 to 3 years, reduce scoliosis, and temper pulmonary and cardiac decline in the second decade of life. However, glucocorticoids causes well-known side effects, which are intolerable in more than 25% of patients. Thus, a disease-specific treatment is a major unmet need. Investigators have proposed various possibilities for the beneficial effects of corticosteroid based mainly on observations in mouse models of muscular dystrophy and on a limited number of studies in patients.

These possibilities include

1. Reducing cytotoxic T lymphocytes
2. Increasing Laminin expression and myogenic repair
3. Retarding muscle apoptosis and cellular infiltration
4. Enhancing Dystrophin expression
5. Affecting neuromuscular transmission

Some patients with Duchenne Myopathy treated early with steroids appear to have an improved long-term prognosis in muscle, myocardial outcome, and can help keep patients ambulatory for more years than expected without treatment. One protocol gives prednisone (0.75 mg/kg/day) for the 1st 10 days of each month to avoid chronic complications. Deflazacort, administered as 0.9 mg/kg/day, may be more effective than prednisone. The American Academy of Neurology and the Child Neurology Society recommend administering corticosteroids during the ambulatory stage of the disease.Published recommendations suggest starting therapy between 2 and 5 years of age in boys whose strength has plateaued or is declining, but earlier treatment may be more beneficial.

Skeletal muscle has a great capacity to regenerate following muscle wasting caused by trauma or disease.This regenerative potential is attributed primarily to skeletal-muscle resident stem cells called satellite cells. In Duchenne Myopathy, satellite cells are exhausted following many rounds of muscle degeneration and regeneration. Hence, satellite cells and their progeny (myoblasts) have been considered as a promising candidate for cell replacement therapy for DMD and other types of muscle disease. Small quantities of adult stem cells exist in most tissues throughout the body where they remain quiescent for long periods of time prior to being activated in response to disease or tissue injury. Adult stem cells can be isolated from cells of the hematopoietic, neural, dermal, muscle and hepatic systems. Adult stem cells give rise to cell types of the tissue from which they originated, but according to scientific reports, they can differentiate into lineages other than their tissue of origin, e.g. transplanted bone marrow or enriched hematopoietic stem cells (HSCs) were reported to give rise to cells of the mesoderm, endoderm and ectoderm.

Two main types of stem cells usually derived from adult bone marrow are HSCs and mesenchymal stem cells (MSC). They can sometimes be obtained from fat, skin, periosteum, synovial membrane and muscle as well. MSCs are multipotent and capable of differentiating into several connective tissue types including osteocytes, chondrocytes, adipocytes, tenocytes and myoblasts. They can also impose an additional anti-inflammatory and paracrine effect on differentiation and tissue regeneration via cytokine pathways and have anti-apoptotic features. These genetically determined pluripotent cells may be easily isolated from bone marrow because they have membrane proteins (marker called cluster of differentiation (CD34 +) and specific marker STRO-I). Compared with pluripotent embryonic stem cells or induced pluripotent stem cells, mesenchymal stem cell have a greater biosafety profile and lower risk of tumorigenicity, and perhaps that is why numerous -mesenchymal stem cell based therapies have made it to the clinical trial stage. Stem cell based therapies for the treatment of Duchenne Myopathy can proceed via two strategies.

The first is autologous stem cell transfer involving cells from a patient with Duchenne Myopathy that are genetically altered in vitro to restore dystrophin expression and are subsequently re-implanted. The second is allogenic stem cell transfer, containing cells from an individual with functional dystrophin, which are transplanted into a dystrophic patient.

Intramuscular route of administration can be considered most appropriate as muscular dystrophy is primarily a muscle disease. The cells can be injected in several points in the muscle alternatively they can be injected in the motor point of the muscle. A motor point is the point at which the motor branch of the innervating nerve enters the muscle. It is the point with the highest concentration of motor endplates and myoneural synapses. Due to high numbers of neuromuscular junctions at this point, a muscle contraction can be easily elicited using minimal electric stimulus. Motor points can therefore be identified as superficial points directly over the points on the muscles with help of external electrical stimulation. Limitation of this method is that only superficial muscles can be stimulated using this method.

In an open study, Sharma and colleagues demonstrated the efficacy of autologous bone marrow mononuclear transplantation by intramuscularly to patients with Duchenne Myopathy, Becker muscular dystrophy and limb girdle muscular dystrophy. However, they did not provide the molecular diagnosis of these dystrophies. No significant adverse events were noted. An increase in trunk muscle strength was seen in 53% of the cases, 48% showed an increase in upper limb strength, 59% showed an increase in lower limb strength and approximately 10% showed improved gait. Eighty seven percent of 150 patients had functional improvement upon physical examination and electromyogram studies after 12 month.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of DMD confirmed by electromyogram (EMG) , Creatine phosphokinase (CPK) level and/ or DNA analysis or muscle biopsy.
* Male patients
* Age 5-15y.
* Ambulatory (loss of ambulation was only seen in those with baseline 6 Minute Walk Distance {6MWD} <325 meters.)
* No clinical evidence of heart failure.

Exclusion Criteria:

* Female patients
* Any injury which may impact functional testing, e.g. upper or lower limb fracture.
* hypertension, diabetes,
* Wheelchair bound.
* Cardiac rhythm disorder, specifically: rhythm other than sinus, supraventricular tachycardia (SVT), atrial fibrillation, ventricular tachycardia.or heart failure (left ventricle ejection fraction {LVEF < 50%}.
* Continuous ventilatory support.
* Liver disease (acute, chronic liver disease)
* Renal impairment

Ages: 5 Years to 15 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — only male
Enrollment: 45 (Estimated)
Dates: Start 2018-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-11 (Estimated)

PRIMARY OUTCOMES:
6 Minute Walk Distance (6MWD) | 6 month
  It is used as measure of motor strength in patients with Duchenne Myopathy. A baseline 6MWD of <350 meters was associated with greater functional decline, and loss of ambulation was only seen in those with baseline 6MWD <325 meters

CONTACTS AND LOCATIONS:
Overall Officials: Emad EL Daly, Professor, Study Director — Assiut University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mercuri E, Muntoni F. Muscular dystrophies. Lancet. 2013 Mar 9;381(9869):845-60. doi: 10.1016/S0140-6736(12)61897-2. PMID 23465426
- [Background] Nallamilli BR, Ankala A, Hegde M. Molecular diagnosis of Duchenne muscular dystrophy. Curr Protoc Hum Genet. 2014 Oct 1;83:9.25.1-29. doi: 10.1002/0471142905.hg0925s83. PMID 25271841
- [Background] Lapidos KA, Kakkar R, McNally EM. The dystrophin glycoprotein complex: signaling strength and integrity for the sarcolemma. Circ Res. 2004 Apr 30;94(8):1023-31. doi: 10.1161/01.RES.0000126574.61061.25. PMID 15117830
- [Background] Emery AE. The muscular dystrophies. Lancet. 2002 Feb 23;359(9307):687-95. doi: 10.1016/S0140-6736(02)07815-7. PMID 11879882
- [Background] Wong BL, Christopher C. Corticosteroids in Duchenne muscular dystrophy: a reappraisal. J Child Neurol. 2002 Mar;17(3):183-90. doi: 10.1177/088307380201700306. PMID 12026233
- [Background] Khan MA. Corticosteroid therapy in Duchenne muscular dystrophy. J Neurol Sci. 1993 Dec 1;120(1):8-14. doi: 10.1016/0022-510x(93)90017-s. PMID 8289083
- [Background] Kojima S, Takagi A, Watanabe T. [Effect of prednisolone on apoptosis and cellular infiltration in mdx mouse muscle]. Rinsho Shinkeigaku. 1999 Nov;39(11):1109-13. Japanese. PMID 10689931
- [Background] Fukudome T, Shibuya N, Yoshimura T, Eguchi K. Short-term effects of prednisolone on neuromuscular transmission in the isolated mdx mouse diaphragm. Tohoku J Exp Med. 2000 Nov;192(3):211-7. doi: 10.1620/tjem.192.211. PMID 11249150
- [Background] Wang YX, Rudnicki MA. Satellite cells, the engines of muscle repair. Nat Rev Mol Cell Biol. 2011 Dec 21;13(2):127-33. doi: 10.1038/nrm3265. PMID 22186952
- [Background] Heslop L, Morgan JE, Partridge TA. Evidence for a myogenic stem cell that is exhausted in dystrophic muscle. J Cell Sci. 2000 Jun;113 ( Pt 12):2299-308. doi: 10.1242/jcs.113.12.2299. PMID 10825301
- [Background] Galli R, Borello U, Gritti A, Minasi MG, Bjornson C, Coletta M, Mora M, De Angelis MG, Fiocco R, Cossu G, Vescovi AL. Skeletal myogenic potential of human and mouse neural stem cells. Nat Neurosci. 2000 Oct;3(10):986-91. doi: 10.1038/79924. PMID 11017170
- [Background] Toma JG, Akhavan M, Fernandes KJ, Barnabe-Heider F, Sadikot A, Kaplan DR, Miller FD. Isolation of multipotent adult stem cells from the dermis of mammalian skin. Nat Cell Biol. 2001 Sep;3(9):778-84. doi: 10.1038/ncb0901-778. PMID 11533656
- [Background] Qu-Petersen Z, Deasy B, Jankowski R, Ikezawa M, Cummins J, Pruchnic R, Mytinger J, Cao B, Gates C, Wernig A, Huard J. Identification of a novel population of muscle stem cells in mice: potential for muscle regeneration. J Cell Biol. 2002 May 27;157(5):851-64. doi: 10.1083/jcb.200108150. Epub 2002 May 20. PMID 12021255
- [Background] Shafritz DA, Oertel M, Menthena A, Nierhoff D, Dabeva MD. Liver stem cells and prospects for liver reconstitution by transplanted cells. Hepatology. 2006 Feb;43(2 Suppl 1):S89-98. doi: 10.1002/hep.21047. PMID 16447292
- [Background] Price FD, Kuroda K, Rudnicki MA. Stem cell based therapies to treat muscular dystrophy. Biochim Biophys Acta. 2007 Feb;1772(2):272-83. doi: 10.1016/j.bbadis.2006.08.011. Epub 2006 Sep 6. PMID 17034994
- [Background] Keating A. Mesenchymal stromal cells: new directions. Cell Stem Cell. 2012 Jun 14;10(6):709-716. doi: 10.1016/j.stem.2012.05.015. PMID 22704511
- [Background] Mendell JR, Clark KR. Challenges for gene therapy for muscular dystrophy. Curr Neurol Neurosci Rep. 2006 Jan;6(1):47-56. doi: 10.1007/s11910-996-0009-8. PMID 16469271
- [Background] Partridge TA. Stem cell therapies for neuromuscular diseases. Acta Neurol Belg. 2004 Dec;104(4):141-7. PMID 15742603